CLINICAL TRIAL: NCT02455908
Title: Use of IL-2 for Pediatric, Multi Drug Resistant, Idiopathic Nephrotic Syndrome
Brief Title: IL-2 for Multi Drug Resistant Nephrotic Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Istituto Giannina Gaslini (Other)
Responsible Party: Principal Investigator, Gian Marco Ghiggeri MD, PhD, MD, director of Nephrology, Dialysis and Transplantation Unit, Istituto Giannina Gaslini
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IL-2 off label
Record Dates: First submitted 2015-05-13; First posted 2015-05-28 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome | interventions — aldesleukin; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Proleukin® (Experimental): Subcutaneous administration of low doses of IL2 (Proleukin) following the therapeutical scheme indicated for crioglobulinemic nephropathy:
  cycle1: IL2 1x106 /m2 s.c for 5 consecutive days cycle2: IL2 1.5 x106 / m2 s.c for 5 consecutive days, starting from 3 weeks after the first cycle.
  cycle3: IL2 1.5 x106 /m2 s.c for 5 consecutive days, starting from 6 weeks after the first cycle.
  Cycle 4: IL2 1.5 x106 /m2 s.c for 5 consecutive days, starting from 9 weeks after the first cycle.
  Interventions: Drug: Proleukin®

INTERVENTIONS:
Drug: Proleukin®
  Other Names: IL-2

SUMMARY:
The aim of the study is to design an open-label phase 1-2 trial to assess safety and clinical and immunologic effects of repeated administration of recombinant low dose IL2 (Proleukin) in 5 patients with idiopathic nephrotic syndrome unresponsive to drugs (steroids, calcineurin inhibitors, Rituximab), following the therapeutical scheme indicated for crioglobulinemic nephropathy:

cycle1: IL2 1x106 /m2 s.c for 5 consecutive days cycle2: IL2 1.5 x106 / m2 s.c for 5 consecutive days, starting from 3 weeks after the first cycle.

cycle3: IL2 1.5 x106 /m2 s.c for 5 consecutive days, starting from 6 weeks after the first cycle.

Cycle 4: IL2 1.5 x106 /m2 s.c for 5 consecutive days, starting from 9 weeks after the first cycle.

Current therapy with steroids and calcineurin inhibitors (Prograf) will be maintained during the first cycle and progressively reduced during the subsequent cycles.

The first cycle will be performed during hospitalization in the investigators Unit; subsequent cycles will be performed at nephrology outpatients. All laboratory values normally utilized in the follow up of patients affected by idiopathic nephrotic syndrome will be evaluated during the first week of treatment and at the end of the protocol, together with specific cellular values (Tregs, B cells, NK).

ELIGIBILITY:
Inclusion Criteria:

* Drug resistance: persistence of proteinuria in nephrotic range after a cycle of steroids of at least 3 months and an association with cyclosporine/tacrolimus for at least other 6 months
* Parents'/guardian's written informed consent, and child's assent given before any study-related procedure not part of the subject's normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to his or her future medical care.
* Age between 2 and 18 years
* Histological pattern of minimal change disease, mesangial proliferation with IgM deposits or focal segmental glomerulosclerosis

Exclusion Criteria:

* Positivity to autoimmunity tests (ANA, dsDNA, ANCA).
* Reduction of C3 levels.
* Hystological pattern characterized by elements suggestive for congenital disease: diffuse mesangial sclerosis without IgM deposits, cystic-like tubular dilatation, mitochondrial abnormalities evident on electron microscopy, IF suggestive for congenital collagen 4 disease.
* Histological pattern not suitable with INS in the pediatric age (membranous glomerulonephritis, lupus nephritis, diffuse and/or localized vasculitis, amyloidosis)
* Homozygous or heterozygous mutations of to the 3 genes (NPHS1, NPHS2, WT1) whose mutations are known to be responsible of almost 80% of familiar cases

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2012-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Proteinuria | Change from baseline at 30, 60 and 180 days after first cycle (5 days)
  Complete remission is defined by urinary protein/creatinine ratio (uPCR) <200 mg/g (<20mg/mmol) for 3 consecutive days. Partial remission is defined as proteinuria reduction of 50% or greater from the presenting value and absolute uPCR between 200 and 2000 mg/g. for 3 consecutive days.

SECONDARY OUTCOMES:
Tregs Levels | Immediately before first cycle and 30, 60 and 180 days after first cycle (5 days)
Serum Creatinine | Change from baseline at 30, 60 and 180 days after first cycle (5 days)
Adverse events | From day 1 to day 5 of each cycle. The study includes 5 cycles, each one lasting 5 days.

CONTACTS AND LOCATIONS:
Overall Officials: Gian Marco Ghiggeri, MD, Principal Investigator — Istituto Giannina Gaslini
Locations (1):
- Istituto Giannina Gaslini, Genova, Italy, Italy

REFERENCES:
- [Background] Trompeter RS, Lloyd BW, Hicks J, White RH, Cameron JS. Long-term outcome for children with minimal-change nephrotic syndrome. Lancet. 1985 Feb 16;1(8425):368-70. doi: 10.1016/s0140-6736(85)91387-x. PMID 2857421
- [Background] Sanna-Cherchi S, Caridi G, Weng PL, Scolari F, Perfumo F, Gharavi AG, Ghiggeri GM. Genetic approaches to human renal agenesis/hypoplasia and dysplasia. Pediatr Nephrol. 2007 Oct;22(10):1675-84. doi: 10.1007/s00467-007-0479-1. Epub 2007 Apr 17. PMID 17437132
- [Background] Pollak MR. Familial FSGS. Adv Chronic Kidney Dis. 2014 Sep;21(5):422-5. doi: 10.1053/j.ackd.2014.06.001. PMID 25168831
- [Background] Vincenti F, Ghiggeri GM. New insights into the pathogenesis and the therapy of recurrent focal glomerulosclerosis. Am J Transplant. 2005 Jun;5(6):1179-85. doi: 10.1111/j.1600-6143.2005.00968.x. PMID 15888021
- [Background] Reiser J, von Gersdorff G, Loos M, Oh J, Asanuma K, Giardino L, Rastaldi MP, Calvaresi N, Watanabe H, Schwarz K, Faul C, Kretzler M, Davidson A, Sugimoto H, Kalluri R, Sharpe AH, Kreidberg JA, Mundel P. Induction of B7-1 in podocytes is associated with nephrotic syndrome. J Clin Invest. 2004 May;113(10):1390-7. doi: 10.1172/JCI20402. PMID 15146236
- [Background] Bertelli R, Bodria M, Nobile M, Alloisio S, Barbieri R, Montobbio G, Patrone P, Ghiggeri GM. Regulation of innate immunity by the nucleotide pathway in children with idiopathic nephrotic syndrome. Clin Exp Immunol. 2011 Oct;166(1):55-63. doi: 10.1111/j.1365-2249.2011.04441.x. Epub 2011 Jul 15. PMID 21762125
- [Background] Ghiggeri GM, Cercignani G, Ginevri F, Bertelli R, Zetta L, Greco F, Candiano G, Trivelli A, Gusmano R. Puromycin aminonucleoside metabolism by glomeruli and glomerular epithelial cells in vitro. Kidney Int. 1991 Jul;40(1):35-42. doi: 10.1038/ki.1991.176. PMID 1921153
- [Background] Ginevri F, Gusmano R, Oleggini R, Acerbo S, Bertelli R, Perfumo F, Cercignani G, Allegrini S, D'Allegri F, Ghiggeri G. Renal purine efflux and xanthine oxidase activity during experimental nephrosis in rats: difference between puromycin aminonucleoside and adriamycin nephrosis. Clin Sci (Lond). 1990 Mar;78(3):283-93. doi: 10.1042/cs0780283. PMID 2156648
- [Background] Garin EH, Diaz LN, Mu W, Wasserfall C, Araya C, Segal M, Johnson RJ. Urinary CD80 excretion increases in idiopathic minimal-change disease. J Am Soc Nephrol. 2009 Feb;20(2):260-6. doi: 10.1681/ASN.2007080836. Epub 2008 Dec 3. PMID 19056875
- [Background] Le Berre L, Bruneau S, Naulet J, Renaudin K, Buzelin F, Usal C, Smit H, Condamine T, Soulillou JP, Dantal J. Induction of T regulatory cells attenuates idiopathic nephrotic syndrome. J Am Soc Nephrol. 2009 Jan;20(1):57-67. doi: 10.1681/ASN.2007111244. Epub 2008 Nov 19. PMID 19020006
- [Background] Wang YM, Zhang GY, Hu M, Polhill T, Sawyer A, Zhou JJ, Saito M, Watson D, Wu H, Wang Y, Wang XM, Wang Y, Harris DC, Alexander SI. CD8+ regulatory T cells induced by T cell vaccination protect against autoimmune nephritis. J Am Soc Nephrol. 2012 Jun;23(6):1058-67. doi: 10.1681/ASN.2011090914. Epub 2012 Apr 5. PMID 22491420
- [Background] Bertelli R, Di Donato A, Cioni M, Grassi F, Ikehata M, Bonanni A, Rastaldi MP, Ghiggeri GM. LPS nephropathy in mice is ameliorated by IL-2 independently of regulatory T cells activity. PLoS One. 2014 Oct 24;9(10):e111285. doi: 10.1371/journal.pone.0111285. eCollection 2014. PMID 25343479
- [Background] Polhill T, Zhang GY, Hu M, Sawyer A, Zhou JJ, Saito M, Webster KE, Wang Y, Wang Y, Grey ST, Sprent J, Harris DC, Alexander SI, Wang YM. IL-2/IL-2Ab complexes induce regulatory T cell expansion and protect against proteinuric CKD. J Am Soc Nephrol. 2012 Aug;23(8):1303-8. doi: 10.1681/ASN.2011111130. Epub 2012 Jun 7. PMID 22677553
- [Background] Saadoun D, Rosenzwajg M, Joly F, Six A, Carrat F, Thibault V, Sene D, Cacoub P, Klatzmann D. Regulatory T-cell responses to low-dose interleukin-2 in HCV-induced vasculitis. N Engl J Med. 2011 Dec 1;365(22):2067-77. doi: 10.1056/NEJMoa1105143. PMID 22129253
- [Background] Koreth J, Matsuoka K, Kim HT, McDonough SM, Bindra B, Alyea EP 3rd, Armand P, Cutler C, Ho VT, Treister NS, Bienfang DC, Prasad S, Tzachanis D, Joyce RM, Avigan DE, Antin JH, Ritz J, Soiffer RJ. Interleukin-2 and regulatory T cells in graft-versus-host disease. N Engl J Med. 2011 Dec 1;365(22):2055-66. doi: 10.1056/NEJMoa1108188. PMID 22129252
- [Background] Bertelli R, Trivelli A, Magnasco A, Cioni M, Bodria M, Carrea A, Montobbio G, Barbano G, Ghiggeri GM. Failure of regulation results in an amplified oxidation burst by neutrophils in children with primary nephrotic syndrome. Clin Exp Immunol. 2010 Jul 1;161(1):151-8. doi: 10.1111/j.1365-2249.2010.04160.x. Epub 2010 May 19. PMID 20491793
- [Background] Boyman O, Kovar M, Rubinstein MP, Surh CD, Sprent J. Selective stimulation of T cell subsets with antibody-cytokine immune complexes. Science. 2006 Mar 31;311(5769):1924-7. doi: 10.1126/science.1122927. Epub 2006 Feb 16. PMID 16484453
- [Background] Kim MG, Koo TY, Yan JJ, Lee E, Han KH, Jeong JC, Ro H, Kim BS, Jo SK, Oh KH, Surh CD, Ahn C, Yang J. IL-2/anti-IL-2 complex attenuates renal ischemia-reperfusion injury through expansion of regulatory T cells. J Am Soc Nephrol. 2013 Oct;24(10):1529-36. doi: 10.1681/ASN.2012080784. Epub 2013 Jul 5. PMID 23833258
- [Background] Ravani P, Magnasco A, Edefonti A, Murer L, Rossi R, Ghio L, Benetti E, Scozzola F, Pasini A, Dallera N, Sica F, Belingheri M, Scolari F, Ghiggeri GM. Short-term effects of rituximab in children with steroid- and calcineurin-dependent nephrotic syndrome: a randomized controlled trial. Clin J Am Soc Nephrol. 2011 Jun;6(6):1308-15. doi: 10.2215/CJN.09421010. Epub 2011 May 12. PMID 21566104
- [Background] Ravani P, Ponticelli A, Siciliano C, Fornoni A, Magnasco A, Sica F, Bodria M, Caridi G, Wei C, Belingheri M, Ghio L, Merscher-Gomez S, Edefonti A, Pasini A, Montini G, Murtas C, Wang X, Muruve D, Vaglio A, Martorana D, Pani A, Scolari F, Reiser J, Ghiggeri GM. Rituximab is a safe and effective long-term treatment for children with steroid and calcineurin inhibitor-dependent idiopathic nephrotic syndrome. Kidney Int. 2013 Nov;84(5):1025-33. doi: 10.1038/ki.2013.211. Epub 2013 Jun 5. PMID 23739238
- [Background] Caridi G, Bertelli R, Di Duca M, Dagnino M, Emma F, Onetti Muda A, Scolari F, Miglietti N, Mazzucco G, Murer L, Carrea A, Massella L, Rizzoni G, Perfumo F, Ghiggeri GM. Broadening the spectrum of diseases related to podocin mutations. J Am Soc Nephrol. 2003 May;14(5):1278-86. doi: 10.1097/01.asn.0000060578.79050.e0. PMID 12707396
- [Background] Caridi G, Perfumo F, Ghiggeri GM. NPHS2 (Podocin) mutations in nephrotic syndrome. Clinical spectrum and fine mechanisms. Pediatr Res. 2005 May;57(5 Pt 2):54R-61R. doi: 10.1203/01.PDR.0000160446.01907.B1. Epub 2005 Apr 6. PMID 15817495
- [Derived] Bonanni A, Bertelli R, Rossi R, Bruschi M, Di Donato A, Ravani P, Ghiggeri GM. A Pilot Study of IL2 in Drug-Resistant Idiopathic Nephrotic Syndrome. PLoS One. 2015 Sep 28;10(9):e0138343. doi: 10.1371/journal.pone.0138343. eCollection 2015. PMID 26413873